CLINICAL TRIAL: NCT03879161
Title: A Percutaneous Ultrasound Device With Needle Guide for Vascular Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired IRB status
Sponsor: Johns Hopkins University (Other)
Collaborators: Perceptive Navigation LLC (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00103043; R42HL093879 (NIH); R44HL093879 (NIH); Z1822 (Other: Other)
Record Dates: First submitted 2019-02-28; First posted 2019-03-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Vascular Access
Keywords: Ultrasound; Femoral Artery; Intra-arterial; Catheterization; Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Arm (Experimental): Study participants will be enrolled in the Device Arm and the Vu-Path™ Device will be used to access the femoral artery for intra-arterial chemoembolization.
  Interventions: Device: Vu-Path™

INTERVENTIONS:
Device: Vu-Path™ — Femoral arterial access in eligible participants will be performed using the Vu-Path™.
  Other Names: Percutaneous Ultrasound Device With Needle Guide

SUMMARY:
This first-in-human pilot study seeks to evaluate the feasibility and safety of using a percutaneous ultrasound device with needle guide for vascular access. Eligible participants will undergo the procedure of transcatheter arterial chemoembolization for primary or metastatic liver cancer, as part of participants' clinical care. The percutaneous ultrasound device with needle guide will be deployed in eligible participants at the beginning of the procedure for guiding a needle inside the femoral artery. Once the needle is inside the artery, then a guide wire is advanced inside the needle and vascular access is successfully obtained.

The study will identify whether this ultrasound-based device with needle guide is helpful for guiding a needle inside the femoral artery.

DETAILED DESCRIPTION:
This NIH Small Business Innovation Research (SBIR)-funded study seeks to test a forward-viewing, ultrasound (US)-based device with needle guide for vascular access.

Access to large arteries is an indispensable step of any trans-arterial catheterization procedure. Surface US-guided vascular cannulation greatly improves first-pass success and reduces complications and is recommended as the preferred technique by numerous specialties and governmental agencies. Surface US-guided cannulation has several key limitations, including dependence on operator skills and experience. Safety and success of vascular access could be vastly improved with a single integrated imaging/interventional device with a small footprint that enables a single-hand operation of the US probe and visualizes the operating needle in real-time.

Reliable and accurate real-time image guidance for vascular access has the potential to appreciably impact public health by enhancing patient safety and convenience, improving procedural accuracy and increasing procedure throughput. Successful implementation has the potential to reduce care and complication costs across millions of vascular access procedures.

Vu-Path™ is a small footprint, US-based device with needle guide. It is a dual-lumen instrument with parallel US imaging and interventional lumens. The forward-viewing US transducer is located at the catheter tip and focused such that the tip of the needle in the interventional lumen, and all proximate structures, are always clearly visualized in real time throughout the procedure.

This is a first-in-human pilot study of the Vu-Path™ device, aiming to its establish clinical feasibility and safety for exemplary use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18 years of age or older at the time of enrollment.
* Participants meeting all medical conditions for percutaneous angiography.
* International Normalized Ratio (INR) <1.3.
* Written informed consent to participate in the study.
* Ability to comply with the requirements of the study procedures.

Exclusion Criteria:

* Fibrous tissue in access path.
* Active skin infection at the point of needle insertion.
* Hemophilia, thrombocytopenia, coagulopathy, or other elevated risk for bleeding or abnormal clotting
* Use of antithrombotic medication.
* For participants taking warfarin or other anticoagulant medication, INR >1.3.
* Participants who cannot tolerate mild sedation.
* Participants with the following laboratory values, unless approved by hematologist: Platelet count <100,000/mL, Activated Partial Thromboplastin Time (APTT) >39 sec or Prothrombin Time (PT) >15 sec
* Pregnancy or lactation
* Patient is unable to comply with requirements of the procedure, i.e. holding breath
* Participation in an investigational trial within 30 days of enrollment.
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder, or any chronic condition that could, in the opinion of the investigator, of interfering with the conduct of the study.
* Participants who are uncooperative or cannot follow instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Device Safety as assessed by number of participants with Minor Bleeding | Within 24 hours from intervention
  Device Safety will be assessed by the number of participants experiencing minor bleeding resulting from vascular puncture. Minor bleeding is defined as either a) bleeding that requires no therapy, or has no consequences or, b) requires nominal therapy, or has no consequence or, c) includes overnight admission for observation only.
Device Safety as assessed by number of participants with Major Bleeding | Within 3 days from intervention
  Device Safety will be assessed by the number of participants experiencing major bleeding. Major bleeding is defined as bleeding that either a) requires therapy and minor hospitalization (25-48 hours) or, b) requires major therapy, unplanned increase in level of care and prolonged hospitalization (> 48 hours), or c) has permanent adverse sequelae or, d) results in death.

SECONDARY OUTCOMES:
Technical accuracy as assessed by number of attempts to reach target site | Within 1 hour from intervention
  Number of attempts to reach target site
Technical accuracy as assessed by percentage of first attempt accesses to target site | Within 1 hour from intervention
  Percentage of first attempt accesses to target site.
Technical efficacy as assessed by procedure time (minutes) | Within 1 hour from intervention
  Procedure time is defined as the total time needed for device procedure.
Technical efficacy as assessed by target access time (minutes) | Within 1 hour from intervention
  Target access time is defined as the total time needed from target visualization to target access.
Technical efficacy as assessed by device usage time (minutes) | Within 1 hour from intervention
  Device usage time is defined as the total time needed for device use.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Liddell, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States